CLINICAL TRIAL: NCT05385146
Title: Effect of Chan-Chuang Qigong With Breathing Meditation on Quality of Life in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ching-I Chang (Other)
Collaborators: Taipei Hospital, Taiwan (Other)
Responsible Party: Sponsor-Investigator, Ching-I Chang, Assistant Professor, Chang Gung University of Science and Technology
Organization: Chang Gung University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCHIRB-10601103
Record Dates: First submitted 2022-04-29; First posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer; Quality of Life; Intraoperative Awareness
MeSH Terms: conditions — Breast Neoplasms; Intraoperative Awareness | interventions — Qigong

STUDY DESIGN:
Intervention Model Description: randomized
Masking Description: patients who signed inform consent are randomized into qigong group and control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- qigong group (Experimental): The qigong group received Chan-Chuang qigong therapy with breathing meditation for 15 weeks.Qigong training program consisted of a warm-up, Chan-Chuang qigong, and breathing meditation. The whole process takes about 20 minutes.The qigong was monitored in terms of muscle elasticity and heart rate variability. After practicing the Chan-Chuang qigong, meditation with breathing was conducted for 10 minutes. In the meanwhile, sit down while relaxing with slow breathing and focus on the present feelings, with brain wave (NeuroSky's, Australia) to monitor and confirm that the eSense (attention and relaxation).
  Interventions: Other: qigong
- control group (No Intervention): those in the control group received usual care during the same study period.

INTERVENTIONS:
Other: qigong — Chan-Chuang qigong with breathing meditation for 15 weeks
  Arms: qigong group

SUMMARY:
The aim of this study was to evaluate the effect of the 15 weeks Chan-Chuang qigong program with breathing meditation on quality of life and interoceptive awareness in patients with breast cancer during chemotherapy.

DETAILED DESCRIPTION:
Cancer is the leading cause of death globally, and breast cancer is the number one threat to women's health worldwide. Chemotherapy is the main adjunctive treatment for breast cancer. However, chemotherapy increasingly being employed in the management of breast cancer patients will cause physical and psychological discomfort as reported. The aim of this study was to evaluate the effect of Chan-Chuang qigong therapy with breathing meditation on quality of life and interoceptive awareness in breast cancer patients. This was a randomized controlled trial. Participants were randomly assigned to the qigong group who received Chan-Chuang qigong therapy with breathing meditation for 15 weeks, and the control group who received routine care. The outcomes were measured by using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) and Multidimensional Assessment of Interoceptive Awareness (MAIA).

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥20
2. diagnosed with breast cancer (stages I and II)
3. before receiving chemotherapy
4. conscious clear to communicate.

Exclusion Criteria:

1. severe cardiopulmonary, liver or kidney dysfunction
2. the original law of qigong cases.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire(EORTC QLQ-C30) scores | baseline, Week 6, Week 15.
  Quality of life was assessed using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30).It consists of 30 items to measure multiple aspects that incorporated five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, and nausea/vomiting), a global health status/QoL scale, and six single common items (dyspnea, loss of appetite, insomnia, constipation, diarrhea, and financial difficulties). The scoring system ranged from 1 (not at all) to 4 (very much). High scores for functional items and low scores for symptoms represent the good QoL.There are two questions for the overall quality of life rating, and the ranking ranged from 1 (very poor) to 7 (excellent).
Change in Multidimensional Assessment of Interoceptive Awareness (MAIA-C) scores | baseline, Week 15
  Interoceptive Awareness was assessed using the Chinese version of the Multidimensional Assessment of Interoceptive Awareness (MAIA-C). which adopts the systematic development of a self-filled questionnaire for the research of experiencing inner perception and the assessment of the physical and mental activity. A total of 32 questions were divided into eight dimensions: Noticing, Not distracting, Not worrying, Attention regulation, Emotional awareness, Self-Regulation, Body listening, and Trusting. The scale asks the individual to answer questions about their inner perception and circle the number that best suits their feelings. The answer options for each question ranged between 0 (never) and 5 (always). The higher scores indicating more positively appraised interoceptive awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang CI, Yeh ML, Liao J. Chan-Chuang qigong with breathing meditation improves quality of life and interoceptive awareness in patients with breast cancer: a randomised controlled trial. Support Care Cancer. 2023 Jan 28;31(2):140. doi: 10.1007/s00520-023-07578-w. PMID 36707489